CLINICAL TRIAL: NCT02217150
Title: The DFINE STAR™ Tumor Ablation Prospective Clinical Series
Brief Title: The STAR Prospective Clinical Series
Acronym: PCS
Status: Completed | Type: Observational
Sponsor: DFINE Inc. (Industry)
Responsible Party: Sponsor
Organization: Merit Medical Systems, Inc. (Industry)
Other Study IDs: PCS; 20130370 (Other: WIRB)
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Metastasis to Vertebral Column

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic Lesions to the spine: Patients over the age of 18 receiving treatment using the DFINE Inc. STAR tumor ablation system for palliation of painful metastases of the spine.

SUMMARY:
Prospective clinical series to gather post tumor ablation clinical outcomes from subjects with painful spinal metastases following targeted radiofrequency ablation (t-RFA) treatment with the STAR™ Tumor Ablation System.

ELIGIBILITY:
Inclusion Criteria:

* The STAR™ Tumor Ablation System is indicated for palliative treatment in spinal procedures by ablation of metastatic malignant lesions in a vertebral body.

Exclusion Criteria:

* The device is contraindicated in subjects with heart pacemakers, or other electronic device implants.
* The device is contraindicated in vertebral body levels C1-7.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with painful spinal metastases following t-RFA with the STAR™ Tumor Ablation System.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Pain | 1 month
  Mean change from baseline in worst pain score per NRPS at one month

SECONDARY OUTCOMES:
Change in Quality of Life | 3 months
  Change from baseline at each visit using Functional Assessment of Cancer Therapy - Bone Pain (FACT-BP)
Change if Quality of Life | 3 months
  Change from baseline at each visit using Functional Assessment of Cancer Therapy (FACT-G7)
Change in Function | 3 months
  Change from baseline at each visit using Modified Oswestry Disability Index (MODI)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Bagla, MD, Principal Investigator — Inova Alexandria Hospital
Locations (8):
- United States (8):
  - Palomar Pomerado Health System, Escondido, California
  - University of Southern California, Los Angeles, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Suburban Hospital, Bethesda, Maryland
  - Austin Radiological Associates, Austin, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Providence Sacred Heart Hospital, Spokane, Washington